CLINICAL TRIAL: NCT04400214
Title: The Food Allergy Superheroes Training (FAST) Program: Increasing Adherence to Food Allergy Safety Guidelines
Brief Title: The Food Allergy Superheroes Training (FAST) Program
Acronym: FAST Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kent State University (Other)
Collaborators: Rhode Island Hospital (Other); University of Memphis (Other)
Responsible Party: Principal Investigator, Christopher Flessner, Associate Professor, Department of Psychological Sciences, Kent State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19-121; 19-118 (Other: Kent State University)
Record Dates: First submitted 2020-05-14; First posted 2020-05-22 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Allergy;Food; Adherence, Treatment; Child, Only
Keywords: Food Allergy; Adherence; Skills training; Child
MeSH Terms: conditions — Food Hypersensitivity; Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: Participants enrolled via the open-trial portion of this study will all receive a 5-session skills training intervention (n = 5 participants). All participants enrolled in the randomized trial portion of this study (n = 50 participants) will be randomly assigned to either a 5-session skills training or 5-session food allergy education intervention
Who Masked: Outcomes Assessor
Masking Description: Independent evaluators will assess pre-, post-, and follow-up naturalistic, food allergy assessment outcomes. These evaluators will have no knowledge as to the intervention participants received via their participation in this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food Allergy Superheroes Training (FAST) Program (Experimental): Participants enrolled in this arm of the study will receive 5, 20 minutes skills training sessions designed to promote adherence to food allergy safety guidelines. These sessions will occur over the period of <2 weeks. All sessions will occur at the PIs laboratory or within the participant's home.
  Interventions: Behavioral: Food Allergy Superheroes Training (FAST) Program
- Food Allergy Knowledge (FAK) Intervention (Active Comparator): Participants enrolled in this arm of the study will receive 5, 20 minutes educational training sessions designed to increase knowledge pertaining to food allergies. These sessions will occur over the period of <2 weeks. All sessions will occur at the PIs laboratory or within the participant's home.
  Interventions: Other: Food Allergy Knowledge Intervention

INTERVENTIONS:
Behavioral: Food Allergy Superheroes Training (FAST) Program — The primary aim of the FAST intervention is to 1) increase the young child's understanding of food allergies (FA) and 2) promote-adherence to FA safety guidelines through active skills training. We will achieve this aim through the use of educational materials (session 1) and a developmentally-tailored skills training intervention (session 2-5). Core components embedded within each skill straining session include instructions, modeling, rehearsal, and reinforcement/corrective feedback. The young child and their parent/caregiver will be present for the entirety of all sessions; however, all intervention materials (i.e., educational content, skills training components) are designed with the young child as the primary focal point of interest. All children will be rewarded with a small toy (<$5 value) at the end of each successfully completed session.
  Other Names: FAST Program
  Arms: Food Allergy Superheroes Training (FAST) Program
Other: Food Allergy Knowledge Intervention — The primary aim of the FAK intervention is to increase the young child's understanding of FAs including prevalence, symptoms, and management strategies among other topics. We will achieve this aim through the use of educational materials targeting knowledge acquisition through a variety of didactic materials made freely available through the Food Allergy Research Education (FARE) website (www.foodallergy.org). More specifically, we will employ information embedded within the "Food Allergy 101" segment of the FARE website. The young child and their parent/caregiver will be present for the entirety of all sessions; however, all intervention materials are designed with the young child as the primary focal point of interest. All children will be rewarded with a small toy (<$5 value) at the end of each successfully completed session. All FAK sessions will occur within the child's home and will include informational handouts relevant to the day's session.
  Other Names: FAK intervention
  Arms: Food Allergy Knowledge (FAK) Intervention

SUMMARY:
Among children with a food allergy, strict avoidance (e.g., elimination of allergenic foods from one's diet) is the only intervention capable of preventing potentially devastating health-related sequelae including anaphylaxis and death. Youths from low-income backgrounds are particularly impacted by food allergies and may be the population most apt to benefit from a brief, portable, and engaging skills-based intervention designed to teach young children the skills needed to remain adherent to food allergy safety guidelines. Data collected as part of the proposed project will lay the groundwork for a line of federally-funded intervention research broadly examining how to promote adherence to food allergy safety guidelines among young children from low-income backgrounds through implementation of a robust, efficient, and portable intervention.

DETAILED DESCRIPTION:
The primary aim of this R21 proposal is to test the efficacy of a 5-session intervention designed to increase adherence to FA safety guidelines among low-income, young children (6-8 years of age) with FAs. This intervention, the Food Allergy Superheroes Training (FAST) Program, will be developed and refined across Phases 1a and 1b to target skills beneficial to promote adherence to FA guidelines (i.e., food avoidance). During Phase 1a, we will recruit a parent-child advisory board to aide in integrating principles of behavioral skills training within the FAST Program manual. We will then examine the initial acceptability and feasibility of the FAST Program in an open trial with 10 low-income, young children with FAs to further refine the intervention's content. During Phase 1b, we will randomize 50 young children with a FA who are from a low-income background to receive either the FAST Program or FA knowledge. We will employ developmentally relevant FA assessments (i.e., child-report, role-play, in situ) before, after, and one-month post-intervention as our primary outcomes. Aim 1: Determine feasibility and acceptability of the FAST intervention. We will evaluate the feasibility and acceptability of this intervention with 60 participants (n=10 in pilot trial [Phase 1a] and n=50 in a preliminary randomized trial [Phase 1b]). Aim 2: Estimate the effect size of the FAST intervention relative to FA knowledge alone. Adherence will be measured via a multi-modal, FA assessment including child-report, role-play, and in situ assessment. This form of naturalistic, FA assessment will be designed to measure the child's behavior (i.e., ingest food, touch or play with food, etc.) in a safe yet realistic manner. This study will contribute to the field's knowledge of efficacious interventions for promoting adherence among young children with FAs.

ELIGIBILITY:
Inclusion Criteria:

* 6-8 years of age.
* Demonstrates a food allergy, based upon parent-report and confirmed diagnosis.
* Family considered low-income (income-to-needs ratio <200% of Department of Health and Human Services Federal Poverty Threshold)
* English as child's primary language
* One English-speaking parent/guardian

Exclusion Criteria:

• Neurodevelopmental disorder (i.e., autism spectrum disorder), cognitive delays, or psychiatric disorder, based upon parent-report.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in in situ food assessment score | pre-intervention to post-intervention (approximately 2 weeks), pre-intervention to one-month follow-up (approximately 6 weeks), post-intervention to one-month follow-up (approximately 4 weeks)
  Designed to provide an objective measure of a child's behavior to an unknown food-item in the real world. Modeled after similar methodology employed in prior skills training research. Study Independent Evaluation (IE) will introduce themselves as a visitor seeking to learn more about working with kids. IE will ask the parent for an empty room to setup their materials. After setup, the child will be asked to complete a simple task (e.g., choose a game or toy to play) whereby the child will come into contact with an unknown food-item (e.g., cookie laying on top of a coloring book). IE will provide minimal response to the child's behavior (e.g., eating food). Child?s response will be coded (see Research Strategy), based upon videotaped assessment made possible via a camera placed in the room. Higher scores (ranging from 0 to 3) indicate greater adherence. Inter-rater reliability will be obtained on 30% of in situ food assessments.
Change in role-play food assessment | pre-intervention to post-intervention (approximately 2 weeks), pre-intervention to one-month follow-up (approximately 6 weeks), post-intervention to one-month follow-up (approximately 4 weeks)
  The role-play assessment will occur immediately following the in situ assessment and is modeled upon similar methodology employed in prior skills training research. The study IE verbally presents the young child with a hypothetical scenario. For example, "Let's pretend that you are in your living room and your mom asks you to pick up your toys. While you are picking up your toys, you find candy. What would you do?" The IE will design each scenario so that the physical layout of the room permits the child to exhibit behavior congruent with the described situation. The child?s response will be coded (see Research Strategy), based upon videotaped assessment made possible via a camera placed in the room. Higher scores (ranging from 0 to 3) indicate greater adherence. Inter-rater reliability will be obtained on 30% of role-play food assessments.
Change in child-report food assessment | pre-intervention to post-intervention (approximately 2 weeks), pre-intervention to one-month follow-up (approximately 6 weeks), post-intervention to one-month follow-up (approximately 4 weeks)
  The child-report food assessment will occur immediately following the role-play assessment. The study IE presents a scenario in which a child finds a food-item (e.g., playing at a friend's home). The IE will ask the child to state what he/she would do, if that situation happened to them. The child's response will be coded (see Research Strategy), based upon videotaped assessment made possible via a camera placed in the room. Higher scores (ranging from 0 to 3) indicate greater adherence. Inter-rater reliability will be obtained on 30% of child-report food assessments.

SECONDARY OUTCOMES:
Food Allergy Knowledge Test (FAKT) | pre-intervention to post-intervention (approximately 2 weeks), pre-intervention to one-month follow-up (approximately 6 weeks), post-intervention to one-month follow-up (approximately 4 weeks)
  The FAKT is a 39 question, parent-report measure designed to assess knowledge about food allergies across five domains: General clinical food allergy knowledge, avoiding exposure, epinephrine auto-injector, anaphylaxis, and symptoms. Questions are multiple choice, true/false, or multiple-item (i.e., indicate whether each item is a symptom of a food allergy) formats. The scale yields a total of 59 items that can be scored. Higher scores indicate a great degree of food allergy knowledge. The scale demonstrates strong internal consistency and construct validity with criterion measures of parent educational status, access to food allergy information, insurance status, and epinephrine use. For purposes of the present study, the FAKT will be used as a process measure designed to ensure that basic educational material is received. Higher scores indicate greater overall food allergy knowledge.
Food Allergy Quality of Life - Parent Burden (FAQL-PB) | pre-intervention to post-intervention (approximately 2 weeks), pre-intervention to one-month follow-up (approximately 6 weeks), post-intervention to one-month follow-up (approximately 4 weeks)
  The FAQL-PB is designed to assess the health-related quality of life among parents of children, 0-12 years of age, with a food allergy. Higher scores indicate greater perceived burden. The scale has demonstrated excellent internal consistency and temporal stability and good construct validity.
Food Allergy Management and Adaptation Scale (FAMAS) | pre-intervention to post-intervention (approximately 2 weeks), pre-intervention to one-month follow-up (approximately 6 weeks), post-intervention to one-month follow-up (approximately 4 weeks)
  The FAMAS is a semi-structured interviewed designed to assess variety of domains related to a family's psychosocial adjustment to a child's food allergy. The interview includes a myriad of subscales related to this broader construct including food allergy knowledge, medication availability, symptoms of food allergy, child and family food avoidance, family and child response readiness, and parent and child anxiety among other domains. Evidence suggests that the FAMAS demonstrates excellent inter-rater reliability and strong construct validity. Higher scores indicate greater overall (better) food allergy management.
Food Allergy Impact Scale (FAIS) | pre-intervention to post-intervention (approximately 2 weeks), pre-intervention to one-month follow-up (approximately 6 weeks), post-intervention to one-month follow-up (approximately 4 weeks)
  The FAIS is a 32-item scale designed to measure the impact of a child's food allergies on day-to-day activities within the home including meal preparation, social activities, etc. Higher scores indicate increasing level of impact on family functioning. Prior research suggests that the FAIS demonstrates adequate internal consistency.

OTHER OUTCOMES:
Child Behavior Checklist (CBCL) | pre-intervention to post-intervention (approximately 2 weeks), pre-intervention to one-month follow-up (approximately 6 weeks), post-intervention to one-month follow-up (approximately 4 weeks)
  The CBCL is a 112-item parent-report scale assessing child symptoms across several domains including social skills, school functioning, and emotional and behavioral problems. Prior research utilizing the CBCL demonstrates strong reliability and validity amongst youth populations. Although multiple versions of the CBCL exist, we will employ the parent-report (6-18 year old) version. For the purposes of the proposed study, we will employ the CBCL as a post hoc measure to assess potential predictors of intervention response. Higher scores on CBCL subscales indicate a greater presence of corresponding behavioral symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Kent State University, Kent, Ohio, United States

REFERENCES:
- See also: PI's laboratory webpage with greater detail about the study and related projects — http://www.ksuparc.org